CLINICAL TRIAL: NCT06258083
Title: Systemic Right Ventricle Long-term Outcome: a Multicentre Study
Brief Title: Systemic Right Ventricle Long-term Outcome
Acronym: SINCERE
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Hartekind (Unknown); Hartstichting (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202100379
Record Dates: First submitted 2023-11-14; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Transposition of the Great Arteries; Systemic Right Ventricle
Keywords: Long-term outcome; Heart failure; Arrhythmias; Mortality
MeSH Terms: conditions — Transposition of Great Vessels; Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Systemic right ventricle patients

SUMMARY:
Patients with the transposition of great arteries (TGA) who undergo atrial switch operation and congenitally corrected TGA (ccTGA) patients have the right ventricle as their systemic ventricle. Function of the systemic right ventricle (SRV) could deteriorate which is associated with impaired prognosis. It is of paramount importance to understand the course and fate of these patients during a long-term follow-up to identify the determinants of adverse outcomes.

DETAILED DESCRIPTION:
In the year 2000, the prevalence of congenital heart diseases (CHD) patients with transposition of great arteries (TGA) was 0.027% in living children and 0.004% in living adults (1). Considering a complete transition to arterial switch operation in the 1990s, it is expected that the number of patients with systemic right ventricle (SRV) decrease over time (2). However, considering the existing number of patients with the TGA who have not undergone arterial switch surgery, SRV remains a challenging issue in the practice of adult congenital heart disease (ACHD) specialists.

TGA is characterized by AV concordance and ventriculo-arterial discordance and is called simple without the presence of associated congenital anomalies. However, complex TGA is when other anomalies are present including VSD (∼45%), LVOTO (∼25%), and CoA (∼5%). TGA's pathogenesis is controversial and there is rare familial occurrence. Male are two times more affected than females. The prognosis of TGA patients without surgery is poor and only exceptional cases survive to adulthood (3).

Heart failure and sudden cardiac death (SCD) are the predominant causes of mortality in TGA patients (4). Patients who undergo atrial switch operation and congenitally corrected TGA (ccTGA) patients are at risk of developing SRV failure in the future (3). The RV is a thin-walled triangular structure acting as a low pressure pump in the normal heart. Because of having only 2 layers, the RV cannot cause the torsion caused by the LV. Due to this geometry and anatomy, the right ventricular function is highly dependent on the loading conditions. The increased afterload that the RV faces in the systemic position causes compensatory RV dilation to maintain the stroke volume. Subsequently, there is increased myocardial wall stress and oxygen demand. The development of heart failure in the SRV is multifactorial. Other potential factors contributing to the SRV failure are impaired coronary reserve or ischemia, myocardial fibrosis, chronotropic incompetence, volume overload from tricuspid regurgitation and arrhythmias (4). Another contributing factor is the reduced baffle compliance in patients with atrial switch. This impairs the preload and stroke volume, especially when there is increased demand. The non-contractile atrial baffles cause impaired atrioventricular transport during tachycardia, therefore causing an inadequate RV filling (4).

Unfortunately, at the moment, the hypothesis that angiotensin-converting enzyme inhibitors (ACE inhibitors), angiotensin II receptor blockers (ARBs), aldosterone antagonists, and beta-blockers can improve the outcome of such patients alone or in combination is not supported by data and evidence. There is no solid recommendation in the 2020 guidelines for the management of ACHD (3).

Previous studies evaluating the fate and outcome of patients with an SRV are either mostly single-centered with a small number of patients or have a short follow-up period (5,6). In a study done by Richard Dobson and colleagues on a national cohort in Scotland, the investigators concluded that patients with an SRV who survive to adulthood have low mortality and good functional status up to the age of 40 (7).

It is of paramount importance to understand the course and fate of these patients during a long-term follow-up to identify the determinants of adverse outcomes. This will enable the investigators to investigate mechanistic pathways of such outcomes. By understanding the risk factors and pathophysiological basis, the investigators can also investigate new diagnostic methods and therapeutic options to improve the quality of life and reduce the mortality of patients with an SRV.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 years old and older
* Surgically corrected transposition of the great arteries (TGA) patients with a systemic right ventricle (SRV) (Mustard, Senning)
* Congenitally corrected TGA patients with a systemic right ventricle

Exclusion Criteria:

* None.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with systemic right ventricles who are followed up in different academic centers in the Netherlands and Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 542 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Through study completion, an average of 18 years
  Death
Incident heart failure | Through study completion, an average of 18 years
  Initiation or increase in dosage (if previously prescribed for another cause, i.e. hypertension) of loop diuretic, ACE-inhibitor/ARB therapy, or evidence-based beta blocker therapy because of new heart failure signs and symptoms (shortness of breath, fatigue, reduced exercise tolerance) AND AT LEAST 1 OF THE FOLLOWING: • BNP ≥400 pg/mL OR the following NT-proBNP levels according to age: < 50 years, ≥450 ng/L; 50-75 years, ≥900 ng/L; >75 years, ≥1800 ng/L OR systolic dysfunction (Systemic ventricle EF <50%) OR • BNP 100-400 pg/mL (or NT-proBNP levels below the thresholds according to age given above) AND structural or functional heart disease
Number of patients with heart failure hospitalization | Through study completion, an average of 18 years
  Rehospitalization, emergency ward visit, 24h observation stay AND Treatment with or increase in dosage if previously prescribed for another cause (i.e.hypertension) of loop diuretics or treatment with IV vasoactive agents.
Number of patients with arrhythmias | Through study completion, an average of 18 years
  Events that cause emergency ward visit or hospitalization.
Number of patients with thromboembolic events | Through study completion, an average of 18 years
  Cerebrovascular events including any of (Hemorrhagic or ischemic): 1, TIA (symptoms less than 24 hours) 2, CVA (symptoms more than 24 hours) and also pulmonary embolism.
Infective endocarditis | Through study completion, an average of 18 years
  Definitie Infective Endocarditis
Number of patients with tricuspid valve surgery | Through study completion, an average of 18 years
  Tricuspid valve surgery
Number of patients with ventricular Assist Device implantation | Through study completion, an average of 18 years
  Implantation of ventricular assist device
Number of patients with heart transplantation | Through study completion, an average of 18 years
  Heart transplantation
Number of patients with aortic aneurysm or dissection | Through study completion, an average of 18 years
  Aortic root more than 40 mm or aneurysm in other parts of aorta. Aortic dissection.
Number of patients with pulmonary artery hypertension | Through study completion, an average of 18 years
  Mean PAP of more than 25mmHg or systolic PAP of more than 40 mmHg.
Number of patients with baffle interventions | Through study completion, an average of 18 years
  Surgical or angiographic reintervention of baffles in patients with surgically corrected transposition of the great arteries (due to stenosis or leakage).
Number of patients with coronary artery interventions | Through study completion, an average of 18 years
  Due to ischemia. Angiographic or surgical intervention.
Number of patients with device implantation | Through study completion, an average of 18 years
  Including pacmakers, ICDs and CRTs.

SECONDARY OUTCOMES:
Number of patients with decreased exercise capacity | At two time points. 1: Baseline 2. Through study completion, an average of 18 years
  Evaluated by cardiopulmonary exercise test results.
Number of patients with right ventricular systolic dysfunction | At two time points. 1: Baseline 2. Through study completion, an average of 18 years
  Measured by echocardiography qualitatively
Number of patients with left ventricular systolic dysfunction | At two time points. 1: Baseline 2. Through study completion, an average of 18 years
  Measured by echocardiography qualitatively

CONTACTS AND LOCATIONS:
Overall Officials: Joost P van Melle, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (9):
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Netherlands (8):
  - Amsterdam University Medical Centre, Amsterdam
  - Medisch Spectrum Twente Enschede, Enschede
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - Maastricht University Medical Centre, Maastricht
  - Radboud University Medical Centre, Nijmegen
  - Erasmus University Medical Centre, Rotterdam
  - University Medical Centre Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marelli AJ, Mackie AS, Ionescu-Ittu R, Rahme E, Pilote L. Congenital heart disease in the general population: changing prevalence and age distribution. Circulation. 2007 Jan 16;115(2):163-72. doi: 10.1161/CIRCULATIONAHA.106.627224. Epub 2007 Jan 8. PMID 17210844
- [Background] Bull C, Yates R, Sarkar D, Deanfield J, de Leval M. Scientific, ethical, and logistical considerations in introducing a new operation: a retrospective cohort study from paediatric cardiac surgery. BMJ. 2000 Apr 29;320(7243):1168-73. doi: 10.1136/bmj.320.7243.1168. PMID 10784538
- [Background] Baumgartner H, De Backer J, Babu-Narayan SV, Budts W, Chessa M, Diller GP, Lung B, Kluin J, Lang IM, Meijboom F, Moons P, Mulder BJM, Oechslin E, Roos-Hesselink JW, Schwerzmann M, Sondergaard L, Zeppenfeld K; ESC Scientific Document Group. 2020 ESC Guidelines for the management of adult congenital heart disease. Eur Heart J. 2021 Feb 11;42(6):563-645. doi: 10.1093/eurheartj/ehaa554. No abstract available. PMID 32860028
- [Background] Andrade L, Carazo M, Wu F, Kim Y, Wilson W. Mechanisms for heart failure in systemic right ventricle. Heart Fail Rev. 2020 Jul;25(4):599-607. doi: 10.1007/s10741-019-09902-1. PMID 31853794
- [Background] Dennis M, Kotchetkova I, Cordina R, Celermajer DS. Long-Term Follow-up of Adults Following the Atrial Switch Operation for Transposition of the Great Arteries - A Contemporary Cohort. Heart Lung Circ. 2018 Aug;27(8):1011-1017. doi: 10.1016/j.hlc.2017.10.008. Epub 2017 Oct 31. PMID 29525133
- [Background] Smood B, Kirklin JK, Pavnica J, Tresler M, Johnson WH Jr, Cleveland DC, Mauchley DC, Dabal RJ. Congenitally Corrected Transposition Presenting in the First Year of Life: Survival and Fate of the Systemic Right Ventricle. World J Pediatr Congenit Heart Surg. 2019 Jan;10(1):42-49. doi: 10.1177/2150135118813125. PMID 30760124
- [Background] Dobson R, Danton M, Nicola W, Hamish W. The natural and unnatural history of the systemic right ventricle in adult survivors. J Thorac Cardiovasc Surg. 2013 Jun;145(6):1493-501; discussion 1501-3. doi: 10.1016/j.jtcvs.2013.02.030. Epub 2013 Mar 13. PMID 23490252